CLINICAL TRIAL: NCT06713070
Title: Pattern of Gait Abnormality As a Predictor for Disease Progression in Dementia
Brief Title: Role of Gait Analysis in Different Type of Dementia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hanan Samwaeil Attia Salib, Resident doctor, Assiut University
Other Study IDs: Gait analysis in dementia
Record Dates: First submitted 2024-06-02; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-10

CONDITIONS: Dementia; Gait Analysis
Keywords: Dementia; Gait analysis; Prognosis
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort 1 (Dementia): The group that will contain the diseased participants (Dementic patients able to walk and perform gait analysis)

SUMMARY:
Aim for the work is the studying of the existence and pattern of gait impairment in pre-dementia and dementia To examine the association between dual decline in gait and cognition

DETAILED DESCRIPTION:
Dementia is a syndrome usually chronic,characterised by progressive global deterioration in intellect, including memory,learning,orientation,comprehension,judgment,gait, and balance

Gait and balance are the product of successful integration of various posture control mechanisms and locomotion.

There are two basic phases in the full cycle of the step Stance phase Swing phase Slow gait speeds are associated with both cognitive decline and greater risk of dementia So, our aim of this work is to study the existence and pattern of gait balance impairment in patients with different types of dementia and comparison with healthy elderly people.

ELIGIBILITY:
Inclusion Criteria:

* patients with pre-dementia,dementia, and dementia diagnosed according to The Vascular Behaviour and Cognitive Disorder (VASCOG) and on medication Criteria attending Assiut University neurology outpatient clinic and internal department

Exclusion Criteria:

* 1 history of clinic manfist cerebrovascular stroke 2 definitely laterization sign 3 severe cognitive imparment MOCA 4 Spinal or orthopaedic problems 5 long-term use or abuse of medication affect cognition or balance 6 clinical evidence of peripheral neuropathy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 30 to 80 yrs old diagnosed with pre-dementia and/or dementia according to the Vascular Behavior and Cognitive Disorder (VASCOG) who are able to perform gait analysis tests
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Analysis and comparison gait analysis in different types of dementia , pre dementia and elderly people | Baseline
  - The studying of the existence and pattern of gait impairment in pre-dementia and dementia and Role and important gait in prediction of disease progression by
  * The new smart insole PODOSmart®, a new tool for gait analysis recording the gait through sensors in foot tabs for 60 seconds and analysing the data.
  * Advanced athactivity of daily living scale (AADLs).
  * Berg balance test (BBT) . Other tools for gait analysis: Dynamic gait index and Figure 8 walk test So, this will study the association between dual decline in gait and cognition with the risk of dementia. And studying of relationship between gait impairment and Cognitive decline in Dementic patients ,which the greater cognitive decline,the greater gait impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Anwer M Ali, Professor, Study Director — Department of Neuropsychiatry in Assuit University Tertiary Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Livingston G, Huntley J, Sommerlad A, Ames D, Ballard C, Banerjee S, Brayne C, Burns A, Cohen-Mansfield J, Cooper C, Costafreda SG, Dias A, Fox N, Gitlin LN, Howard R, Kales HC, Kivimaki M, Larson EB, Ogunniyi A, Orgeta V, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care: 2020 report of the Lancet Commission. Lancet. 2020 Aug 8;396(10248):413-446. doi: 10.1016/S0140-6736(20)30367-6. Epub 2020 Jul 30. No abstract available. PMID 32738937
- [Background] Jack CR Jr, Knopman DS, Jagust WJ, Petersen RC, Weiner MW, Aisen PS, Shaw LM, Vemuri P, Wiste HJ, Weigand SD, Lesnick TG, Pankratz VS, Donohue MC, Trojanowski JQ. Tracking pathophysiological processes in Alzheimer's disease: an updated hypothetical model of dynamic biomarkers. Lancet Neurol. 2013 Feb;12(2):207-16. doi: 10.1016/S1474-4422(12)70291-0. PMID 23332364
- [Background] Borson S, Raskind MA. Clinical features and pharmacologic treatment of behavioral symptoms of Alzheimer's disease. Neurology. 1997 May;48(5 Suppl 6):S17-24. doi: 10.1212/wnl.48.5_suppl_6.17s. PMID 9153156
- [Background] Rodriguez Garcia PL, Rodriguez Garcia D. Diagnosis of vascular cognitive impairment and its main categories. Neurologia. 2015 May;30(4):223-39. doi: 10.1016/j.nrl.2011.12.014. Epub 2012 Jun 26. English, Spanish. PMID 22739039
- [Background] Dicharry J. Kinematics and kinetics of gait: from lab to clinic. Clin Sports Med. 2010 Jul;29(3):347-64. doi: 10.1016/j.csm.2010.03.013. PMID 20610026
- [Background] Jayakody O, Breslin M, Srikanth VK, Callisaya ML. Gait Characteristics and Cognitive Decline: A Longitudinal Population-Based Study. J Alzheimers Dis. 2019;71(s1):S5-S14. doi: 10.3233/JAD-181157. PMID 30958358
- [Background] Verghese J, Wang C, Lipton RB, Holtzer R, Xue X. Quantitative gait dysfunction and risk of cognitive decline and dementia. J Neurol Neurosurg Psychiatry. 2007 Sep;78(9):929-35. doi: 10.1136/jnnp.2006.106914. Epub 2007 Jan 19. PMID 17237140
- [Background] Moran C, Beare R, Phan TG, Bruce DG, Callisaya ML, Srikanth V; Alzheimer's Disease Neuroimaging Initiative (ADNI). Type 2 diabetes mellitus and biomarkers of neurodegeneration. Neurology. 2015 Sep 29;85(13):1123-30. doi: 10.1212/WNL.0000000000001982. Epub 2015 Sep 2. PMID 26333802
- [Background] Brach JS, Talkowski JB, Strotmeyer ES, Newman AB. Diabetes mellitus and gait dysfunction: possible explanatory factors. Phys Ther. 2008 Nov;88(11):1365-74. doi: 10.2522/ptj.20080016. Epub 2008 Sep 18. PMID 18801861
- [Background] Blumen HM, Brown LL, Habeck C, Allali G, Ayers E, Beauchet O, Callisaya M, Lipton RB, Mathuranath PS, Phan TG, Pradeep Kumar VG, Srikanth V, Verghese J. Gray matter volume covariance patterns associated with gait speed in older adults: a multi-cohort MRI study. Brain Imaging Behav. 2019 Apr;13(2):446-460. doi: 10.1007/s11682-018-9871-7. PMID 29629501
- [Background] Jayakody O, Breslin M, Beare R, Srikanth VK, Blumen HM, Callisaya ML. The Associations Between Grey Matter Volume Covariance Patterns and Gait Variability-The Tasmanian Study of Cognition and Gait. Brain Topogr. 2021 Jul;34(4):478-488. doi: 10.1007/s10548-021-00841-5. Epub 2021 Apr 29. PMID 33914190
- [Background] Rosano C, Studenski SA, Aizenstein HJ, Boudreau RM, Longstreth WT Jr, Newman AB. Slower gait, slower information processing and smaller prefrontal area in older adults. Age Ageing. 2012 Jan;41(1):58-64. doi: 10.1093/ageing/afr113. Epub 2011 Sep 28. PMID 21965414
- [Background] Srikanth V, Beare R, Blizzard L, Phan T, Stapleton J, Chen J, Callisaya M, Martin K, Reutens D. Cerebral white matter lesions, gait, and the risk of incident falls: a prospective population-based study. Stroke. 2009 Jan;40(1):175-80. doi: 10.1161/STROKEAHA.108.524355. Epub 2008 Oct 16. PMID 18927448
- [Background] Del Campo N, Payoux P, Djilali A, Delrieu J, Hoogendijk EO, Rolland Y, Cesari M, Weiner MW, Andrieu S, Vellas B; MAPT/DSA Study Group. Relationship of regional brain beta-amyloid to gait speed. Neurology. 2016 Jan 5;86(1):36-43. doi: 10.1212/WNL.0000000000002235. Epub 2015 Dec 7. PMID 26643548
- [Background] Dias EN, da Silva JV, Pais-Ribeiro JL, Martins T. Validation of the advanced activities of daily living scale. Geriatr Nurs. 2019 Jan-Feb;40(1):7-12. doi: 10.1016/j.gerinurse.2018.05.008. Epub 2018 Jun 13. PMID 29909023
- [Background] Rahman TT, El Gaafary MM. Montreal Cognitive Assessment Arabic version: reliability and validity prevalence of mild cognitive impairment among elderly attending geriatric clubs in Cairo. Geriatr Gerontol Int. 2009 Mar;9(1):54-61. doi: 10.1111/j.1447-0594.2008.00509.x. PMID 19260980
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055